CLINICAL TRIAL: NCT05726201
Title: Point-Of-Care Ultrasound (POCUS) As an Early Screening Tool for Diagnosing Skull Fractures In Children With Mild Closed Head Injuries
Brief Title: (POCUS) As an Early Screening Tool for Diagnosing Skull Fractures in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Professor of Anesthesiology and Intensive Care Faculty of Medicine, Assiut University
Other Study IDs: POCUS for skull fracture
Record Dates: First submitted 2023-01-31; First posted 2023-02-13 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Trauma, Brain
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound — Point-Of-Care Ultrasound (POCUS) As an Early Screening Tool for Diagnosing Skull Fractures In Children With Mild Closed Head Injuries

SUMMARY:
This study aims to evaluate the accuracy of POCUS as a screening tool for early diagnosis of skull fractures in children with mild closed head injuries admitted to the emergency department. The results would aid the emergency physicians to speed up the management and reduce the cost of diagnosing skull fractures and TBI.

DETAILED DESCRIPTION:
Trauma is defined as a physical injury from an external source. Despite improvements in trauma systems worldwide, trauma continues to be one of the leading causes of death and disability in all age groups, especially the young and middle age groups.Head trauma can result in skull fractures which are a common cause of morbidity and mortality in children. There is a high flow of presentations in the Pediatric Emergency Department (PED) and primary care. Children are more susceptible to head trauma and skull fractures than adults. The child's head size is approximately 18% of the total body surface area in infancy. Compared to an adult skull, the child's skull is thinner and more pliable, thus providing less protection to the brain. The Centers for Disease Control and Prevention in the USA reported 749,000 ED visits for injury to the head in children under the age of 15 years old in 2016. One Up to 8% of children aged 3-17.

The Causes of head injury and skull fractures can be classified into accidental and non accidental injuries. Commonly, head injuries are caused by a fall. Other causes can include motor vehicle accidents (MVA), sports-related injuries, or other direct blows to the head. Occasionally, depressed "ping-pong" fractures can occur in newborns due to injury at birth. Fortunately, the majority (80% to 90%) of head injuries can be classified as mild. Very few injuries are life-threatening or require neurosurgical intervention. The incidence of skull fractures in children following head injury ranges from 2% to 20%, and further epidemiological studies are needed for more accurate incidence and prevalence rates.

Skull fractures are more common in children under the age of 2 years following head trauma. A fracture of the calvarium (skull cap) is more common than one at the base of the skull. Skull fractures can cause many complications, such as skin damage, soft tissue injuries, bone fractures, and brain tissue injuries, which are known as traumatic brain injuries. Traumatic brain injury (TBI), which is defined as a disruption in the normal brain's function, can involve both adults and children, but its pathophysiology and management are different in children.

When the skull is fractured, the dura mater is prone to damage. The dural laceration is common in Diastatic skull fractures and should be diagnosed because of its complications.

Head CT scan, an X-ray-based modality, is widely used to diagnose skull fractures and TBI. Children are more sensitive to ionizing radiation, and the relative risk of cancer is higher in them. Identification of skull fractures in children is clinically relevant because these fractures may need surgical intervention irrespective of the presence of TBI. Skull fractures could be associated with non-accidental trauma, and physicians should always consider this potential association .In addition, skull fractures may need follow-up because linear fractures may predispose children to uncommon but serious complications such as expanding fractures or leptomeningeal cysts. Clinicians must weigh the risk of missing a clinically important skull fracture and potentially associated TBI and the risks associated with performing a CT (i.e., carcinogenic effect, and changes in the cognitive function afterwards).

Given the dangers of using X-rays and computed tomography (CT) scans, physicians are attempting to reduce the use of these methods as much as possible. Solutions include the development of clinical guidelines to reduce unnecessary exposure (e.g, PECARN Rule) or alternative imaging methods such as magnetic resonance imaging (MRI) or ultrasonography (US). US is a noninvasive tool that is superior to CT and MRI for detecting dura's status. Also, it is preferred over MRI as being more available in the emergency department.Rabiner et al. stated the following benefits of point-of-care ultrasound (POCUS): (a) early diagnosis of a patient and early consultation; (b) reduction in CT scan request; (c) as a diagnostic tool when there is no access to CT scan; and (d) a triage tool in a disaster area with difficult conditions.Weinberg et al. reported that the accuracy of POCUS was higher in diagnosing longitudinal bone fractures, especially in young adults and children. Recent studies reported high sensitivity and specificity of POCUS in the clinical diagnosis of skull fractures (91%,96% respectively ). It is noticeable that POCUS may be a tool for detecting skull fractures; it does not rule out brain lesions which might be more hazardous for the injured patients, and in high-risk patients, a CT scan should be performed. Although POCUS is considered a good diagnostic tool, extensive use of ultrasound to diagnose skull fractures has significant limitations. Firstly, the location of the injury has to be clearly identified; the skin mustn't have any damage. In many cases, finding the injury location is challenging. Second, is the need for sedation in children to perform this procedure. The need for relaxation and immobility is always one of the challenges of performing ultrasound in children.

The algorithm of the PECARN rule is widely used to decide on performing CT scans in childrenwith mild head trauma . In this algorithm, the use of CT for children with a moderate risk for brain injury has always been challenged, especially when the child visits an ED center where there is no CT scan, and the physician wants to refer the child to a higher-levelcenter for CT. In this case, if the child is eligible for ultrasound, the location of the injury is clear, and the skin is not torn, ultrasound can be used to determine the existence of a skull fracture which would be an indication to perform CT to discard intracranial injuries A recent meta-analysis recommended the consideration of POCUS in patients that meet no other major or multiple minor criteria for a CT scan than a clinically suspected skull fracture, or when a skull fracture cannot be excluded; consequently, when no fracture is identified, a CT scan might not be needed. Therefore, using POCUS to rule out a skull fracture could potentially reduce the utilization of CT and unnecessary exposure of children to ionizing radiation. The aim of POCUS is not to detect TBI, but it can identify skull fracture which is an important predictor of Clinically important TBI (ciTBI).Based on these assumptions, the POCUS is better included in the early screening of children with mild closed head injuries rather than to be a definitive diagnostic tool. This study will screen pediatric patients with mild closed head injury aiming to define the role of POCUS in risk stratification for TBI and its applicability in conjunction with the clinical prediction rules. Thereby, the decision to ''recommend CT'' will be based on both early admission POCUS and PECARN rule.

ELIGIBILITY:
Inclusion Criteria:

* Age group 2 - 18 years old
* Both genders
* Blunt head trauma within 24hours of admission to the ED.
* Glasgow Coma Scale scores of 14 to 15.
* Localizing evidence of scalp trauma (cephalohematoma, focal pain, deformity)

Exclusion Criteria:

* Patients who are less than 2 years old or more than 18 years old
* Patients with open head wounds
* Ventricular shunts
* Bleeding disorders
* Known brain tumors
* Pre-existing neurological disorders complicating assessment

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Age group 2 - 18 years old
  * Both genders
  * Blunt head trauma within 24hours of admission to the ED.
  * Glasgow Coma Scale scores of 14 to 15.
  * Localizing evidence of scalp trauma (cephalohematoma, focal pain, deformity)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-07-23 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
main | 3 years
  Evaluate the diagnostic accuracy (sensitivity and specificity) of point of-care ultrasound (POCUS) as a screening tool for identifying and early diagnosis skull fractures in children with mild closed head trauma

SECONDARY OUTCOMES:
Incidence | 3 years
  Describing the incidence of skull fracture in children
PECARN predictive rule | 3 years
  PECARN predictive rule
Computed Tomography Scanning skull | 3 years
  CT skull findings.
Agreement ratio | 3 years
  the agreement ratio between the results of the POCUS, PECARN rule and CT findings.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assiut University; Zeinab M Abd-Elatiff, MD, Principal Investigator — Suez Canal University
Locations (1):
- Omar Ibrahim Abdelsalam, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided